CLINICAL TRIAL: NCT01510951
Title: A Randomized, Double-blind, Placebo-controlled, Single-dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Clinical Effects of AMG 811 in Subjects With Moderate to Severe Psoriasis
Brief Title: Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Clinical Effects of AMG 811 in Subjects With Psoriasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 20101147
Record Dates: First submitted 2011-08-11; First posted 2012-01-18 (Estimated); Last update posted 2013-03-27 (Estimated); Status verified 2013-03

CONDITIONS: Psoriasis
Keywords: AMGEN; PSORIASIS; SAFETY
MeSH Terms: conditions — Psoriasis | interventions — AMG 811

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- PLACEBO (Placebo Comparator)
  Interventions: Drug: AMG 811 or Placebo
- AMG 811 (Experimental)
  Interventions: Drug: AMG 811 or Placebo

INTERVENTIONS:
Drug: AMG 811 or Placebo — Single dose subcutaneous administration of AMG 811 or placebo to adult subjects with psoriasis.

SUMMARY:
The purpose of this study is to assess the safety, tolerability, immunogenicity, and clinical effects of AMG 811 following single subcutaneous dose administration in subjects with moderate to severe psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 55 years old inclusive at Screening
* Active but clinically stable, plaque psoriasis
* Psoriasis involving ≥ 10% of the body surface area
* A minimum PASI score of ≥ 10 obtained during the screening period
* Additional inclusion criteria apply

Exclusion Criteria:

* Active guttate, erythrodermic, or pustular psoriasis at the time of the screening visit
* Evidence of skin conditions other than psoriasis (eg, eczema) at the time of the screening visit or between the screening visit and study drug initiation that would interfere with evaluations of the effect of investigational product on psoriasis
* Any condition that, in the judgment of the investigator, might cause this study to be detrimental to the subject
* Additional exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2011-08; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Evaluate the number of adverse events per subject, including clinically significant changes in physical examinations, safety lab tests, ECG, vital signs, or immunogenicity to AMG 811 | 16 weeks

SECONDARY OUTCOMES:
Evaluate the efficacy of AMG 811 as measured by the following: the proportion of subjects with a PASI 50, 75 and 90 | 16 weeks
Measure the area under the serum concentration curve versus time of AMG 811 after a single dose administration in subjects with moderate to severe psoriasis | 16 weeks
Measure the peak serum concentration (Cmax) of AMG 811 after a single dose administration in subjects with moderate to severe psoriasis | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (4):
- Australia (2):
  - Research Site, Herston, Queensland
  - Research Site, Nedlands, Western Australia
- New Zealand (2):
  - Research Site, Christchurch
  - Research Site, Grafton, Auckland

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com